CLINICAL TRIAL: NCT07176325
Title: Gastrointestinal and Fluid Retention Symptoms Associated With Creatine Monohydrate With and Without Loading Dose Over 28 Days of Supplementation
Status: Completed | Type: Observational
Sponsor: Vireo Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VIRUSE1R
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Side Effects of Creatine Monohydrate Dosing
Keywords: creatine monohydrate, gastrointestinal symptoms, supplementation, dosing regimen, tolerability, compliance, loading dose
MeSH Terms: conditions — Patient Compliance | interventions — Creatine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A (5 g/day CM): No Loading Group
  Interventions: Other: Creatine Monohydrate
- Group B (20 g/day loading dose for 14 days followed by 5 g/day maintenance): Loading Group
  Interventions: Other: Creatine Monohydrate

INTERVENTIONS:
Other: Creatine Monohydrate — Creatine Monohydrate was dosed based on industry recommendations, with and without a loading dose

SUMMARY:
This study aimed to investigate the incidence and severity of GI symptoms associated with daily CM supplementation, with and without a loading phase, in healthy male and female adults.

DETAILED DESCRIPTION:
In a 28-day single-center, single-blind, randomized clinical trial, 24 healthy participants were assigned to either Group A (5 g/day CM) or Group B (20 g/day loading dose for 14 days followed by 5 g/day maintenance). Blood and urine samples were collected at baseline and day 28 to assess safety. GI symptoms were recorded via self-report using a structured severity rating scale.

ELIGIBILITY:
Inclusion Criteria:

* ○ Subjects must be healthy males or females, aged 18 to 60 inclusive at the time of screening.

  * Subjects must be able to understand the study, agree to the requirements and restrictions, and be willing to give voluntary consent to participate in the study.
  * Subjects are willing to have up to two (2) blood collections, one at Visit 2 and Visit 3.
  * Subjects are willing to provide a urine sample that is collected over 24 hours. This entails collecting all urine in a 24-hour period in a container.
  * Subject is willing to fast for 12 hours before the Baseline visit (second visit). Water is permitted.
  * Subject is willing to have waist measurements taken with calipers and willing to wear clothing that allows easy access to their waist.
  * Female subjects of childbearing potential must agree to one of the following methods of birth control through the duration of the study. Acceptable methods include: abstinence, same-sex partner, double barrier (condom, diaphragm, or cervical cap with spermicidal foam, gel, or cream); intra-uterine device (IUD) with or without hormones in place or hormonal contraception (oral, injectable, implantable, transdermal, or vaginal) used consecutively for at least 3 month prior to screening visit; vasectomized partner or bilateral insertion of Essure® implants (or analogous) for at least 6 months prior to the screening visit; to be considered a female of non- childbearing potential, subject must have had a bilateral tubal ligation, hysterectomy or bilateral oophorectomy; or postmenopausal status with amenorrhea (no menstruation) for at least 1 year prior to the screening visit.
  * Subject is willing to comply with the study restrictions.
  * Subjects is willing to maintain their current exercise regimen and their current diet while on the study.

Exclusion Criteria:

* ○ Subjects who are participating in another Clinical Trial.

  * Subjects who faint during blood collection, or who have a phobia of needles, or a phobia of blood.
  * Subjects who are weightlifters.
  * Females who are pregnant or lactating (verbal confirmation only).
  * Subject who has taken any creatine supplements in the last 30 days.
  * Subjects with history of cancer (except localized skin cancer without metastases) within 5 years prior to the screening visit.
  * Subject has diabetes (insulin dependent or not) or any immune deficiency disease such as HIV/AIDS, etc.
  * Subject has any medical condition whether treating with mediation or not including hypertension (high blood pressure), hepatitis, any kidney disease or disorders, or musculoskeletal disorders. Note: if there are any significantly abnormal results for the BUN/creatinine screening labs the subject will be dropped.
  * Subject is taking a medication that would preclude participation in the study per the Principal Investigator.
  * Subjects with recent or current medical condition that may significantly impact the subject or the validity of the study results in the opinion of the Investigator.
  * Subjects who have a known or suspected allergy or sensitivity to creatine.
  * Chronic use of NSAIDs (e.g., Ibuprofen, Advil), or use of NSAIDs at one-week prior to each study visit.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy male and females ages 18-60
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal distress | 28 days
  Gastrointestinal effects are well known, particularly at higher doses.

CONTACTS AND LOCATIONS:
Locations (1):
- Princeton Consumer Research, Raritan, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We are looking at aggregate trends in the data